CLINICAL TRIAL: NCT03621540
Title: Augmentation of Working Memory Training With Transcranial Direct Current Stimulation (tDCS) in Patients With Schizophrenia
Brief Title: Augmentation of Working Memory Training With Transcranial Direct Current Stimulation in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: ESPRIT Training
Record Dates: First submitted 2018-05-08; First posted 2018-08-08 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Schizophrenia; Cognitive Deficits
Keywords: transcranial direct current stimulation; schizophrenia; cognitive deficits; working memory training
MeSH Terms: conditions — Schizophrenia; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Use of NeuroConn Stimulator study mode
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum arm (Active Comparator): 25 min anodal tDCS + adaptive working memory training
  Interventions: Device: active tDCS; Behavioral: Adaptive working memory training
- Sham arm (Sham Comparator): sham tDCS + adaptive working memory training
  Interventions: Device: sham tDCS; Behavioral: Adaptive working memory training

INTERVENTIONS:
Device: active tDCS — Using the NeuroConn Plus tDCS device, 2 mA anodal tDCS will be applied to the right dorsolateral prefrontal cortex (F4). 15 s fade in and fade out. Total stimulation time of 1365 s. Cathode over contralateral deltoid muscle.
  Arms: Verum arm
Device: sham tDCS — Sham mode of the NeuroConn Plus tDCS device with 2 mA stimulation for 45 s at the beginning. Anode over right dorsolateral prefrontal cortex (F4), Cathode over contralateral deltoid muscle. After that, only continuous impedance checking is performed.
  Arms: Sham arm
Behavioral: Adaptive working memory training — Adaptive spatial n-back training.

SUMMARY:
Cognitive impairment is a core symptom of schizophrenia and is in a large part responsible for the poor psychosocial outcome of the disorder. The use of non-invasive brain stimulation techniques as a therapeutic option is just commencing for neuropsychiatric patients. Concerning healthy subjects the investigators have previously shown that anodal tDCS to the right dorsolateral prefrontal cortex (DLPFC) parallel to working memory training can sustainingly enhance performance in a spatial n-back task. Additionally, first translational experiments regarding the use of anodal tDCS to improve working memory (WM) in patients with schizophrenia rendered promising results.

On those grounds, the investigators now test the hypothesis that anodal tDCS to the right DLPFC can augment working memory training in patients with schizophrenia.

DETAILED DESCRIPTION:
Cognitive impairments are a core and debilitating feature of schizophrenia, but effective treatment options are scarce. These deficits develop early in the progression of the disorder, frequently persist throughout lifespan and are considered a possible endophenotype of the disorder. Everyday functioning, work ability and social integration are substantially affected. A proper treatment of cognitive symptoms would probably reduce individual consequences like unemployment or early retirement and alleviate the resulting cost for our societies.

Working memory, the ability to temporally maintain and manipulate information, is critically relevant as interface between sensory input and the attainment of behavioral goals. It plays a pivotal role in executive functioning and shares overlapping cognitive processes with social cognition. The characteristic WM deficits in patients with schizophrenia are associated with aberrant dlPFC activation and connectivity, rendering this brain region a prime target for treatment interventions. Cognitive and specifically WM training have been proven effective to change prefrontal activation pattern resulting in improved performance. However, the effect sizes are moderate and the expenditure is high, so that training paradigms are not consistently implemented in regular treatment.

A possible way to increase the efficacy of WM training is the augmentation with non-invasive brain stimulation techniques. Transcranial direct current stimulation modulates neuronal membrane potentials and is regulating cortical excitability depending on polarity. Specifically, anodal stimulation can induce long-lasting cortical excitability elevations.

First translational studies exploring the effectiveness of tDCS to enhance cognition in patients with schizophrenia yielded promising results.To extend this knowledge, the investigators examine the effect of a tDCS augmented WM training (2 mA to the right dlPFC) in patients with schizophrenia. The WM training consists of two weeks (10 daily sessions) of 20 minute adaptive spatial n-back training, complemented by a Pre/Post session and two follow-up measurements after 4 and 12 weeks. In the two arms parallel study design, patients will be randomized either to the group receiving active anodal tDCS during the training or to the other group receiving sham stimulation during the training. The investigators hypothesize an enhancement of WM performance by anodal tDCS and investigate possible transfer effects in other cognitive tasks, psychopathology, quality of life and subjective cognitive capabilities. The investigators will further analyze the influence of the genetic make-up, neurophysiological signatures and other demographic and cognitive variables on the stimulation effect.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia or schizoaffective disorder
* age 18-60 years
* Ability to give informed consent
* right handedness
* stable antipsychotic medication one week prior to the experiment and during the training sessions

Exclusion Criteria:

* epilepsy
* metal implants near the head
* pregnancy
* use of antiepileptics
* use of benzodiazepines > 1 mg lorazepam equivalent
* current substance abuse (excluding tabacco)
* missing consent of the legal representative, if existing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Change (post training - pre training) in working memory task performance (1-,2-,3-back). | Pre Training: 3-4 days before training start. Post Training: 3-4 days after completion of working memory training.
  Use of d' and response time as dependent variables. Based on signal detection theory, the discriminability index d' (d-prime) is calculated by using the formula d' = Z(hit rate) - Z(false alarm rate).

SECONDARY OUTCOMES:
Change (post training - pre training) in cognitive flexibility and processing speed. | Pre Training: 3-4 days before training start. Post Training: 3-4 days after completion of training. And changes in follow-up sessions: 4 and 12 weeks after completion of working memory training.
  Trail Making Test (TMT) A and B. Results in seconds will be normalized by age and education adjusted standard values. Slower processing time indicates less cognitive flexibility and processing speed.
Change (follow-up - pre training) in cognitive flexibility and processing speed. | Pre Training: 3-4 days before training start. Follow-up sessions: 4 and 12 weeks after completion of working memory training.
  Trail Making Test (TMT) A and B. Results in seconds will be normalized by age and education adjusted standard values. Slower processing time indicates less cognitive flexibility and processing speed.
Change (post training - pre training) in cognition. | Pre Training: 3-4 days before training start. Post Training: 3-4 days after completion of training. And changes in follow-up sessions: 4 and 12 weeks after completion of working memory training.
  Measure of different cognitive domains with the Brief Assessment of Cognition in Schizophrenia (BACS). Subscales (Verbal Memory, Working Memory, Motor Function, Verbal Fluency, Speed of Processing, Executive Function) and composite score. Taking age and gender into account, individual test scores are averaged to standardized scores (z-score) . Higher scores indicate better task performance.
Change (follow-up - pre training) in cognition. | Pre Training: 3-4 days before training start. Follow-up sessions: 4 and 12 weeks after completion of working memory training.
  Measure of different cognitive domains with the Brief Assessment of Cognition in Schizophrenia (BACS). Subscales (Verbal Memory, Working Memory, Motor Function, Verbal Fluency, Speed of Processing, Executive Function) and composite score. Taking age and gender into account, individual test scores are averaged to standardized scores (z-score) . Higher scores indicate better task performance.
Change (follow-up - pre training) in working memory task performance (1-,2-,3-back). | Pre Training: 3-4 days before training start. Follow up: 4 and 12 weeks after completion of working memory training.
  Use of the d' and response time as dependent variables. Based on signal detection theory, the discriminability index d' (d-prime) is calculated by using the formula d' = Z(hit rate) - Z(false alarm rate).
Change (post training - pre training) in depressive symptoms. | Pre Training: 3-4 days before training start. Post Training: 3-4 days after completion of training.
  Calgary Depression Scale for Schizophrenia (CDSS). Maximum score is 27. Higher scores indicate a higher level of depression.
Change (follow-up - pre training) in depressive symptoms. | Pre Training: 3-4 days before training start. Follow-up sessions: 4 and 12 weeks after completion of working memory training.
  Calgary Depression Scale for Schizophrenia (CDSS). Maximum score is 27. Higher scores indicate a higher level of depression.
Change (post training - pre training) in psychopathology. | Pre Training: 3-4 days before training start. Post Training: 3-4 days after completion of training. And changes in follow-up sessions: 4 and 12 weeks after completion of working memory training.
  Positive and Negative Syndrome Scale (PANSS). The PANSS measures symptom severity on a positive, a negative and a general psychopathology scale. Higher scores indicate more pronounced symptom severity. The PANSS will be analyzed in subscales and as a summed total score.
Change (follow-up - pre training) in psychopathology. | Pre Training: 3-4 days before training start. Follow-up sessions: 4 and 12 weeks after completion of working memory training.
  Positive and Negative Syndrome Scale (PANSS). The PANSS measures symptom severity on a positive, a negative and a general psychopathology scale. Higher scores indicate more pronounced symptom severity. The PANSS will be analyzed in subscales and as a summed total score.
Change (post training - pre training) in negative symptoms | Pre Training: 3-4 days before training start. Post Training: 3-4 days after completion of training.
  Scale for the Assessment of Negative Symptoms (SANS). The total score is calculated by addition of 5 subscales with a maximum score of 25. A higher score indicates more pronounced negative symptoms.
Change (follow-up - pre training) in negative symptoms | Pre Training: 3-4 days before training start. And changes in follow-up sessions: 4 and 12 weeks after completion of working memory training.
  Scale for the Assessment of Negative Symptoms (SANS). The total score is calculated by addition of 5 subscales with a maximum score of 25. A higher score indicates more pronounced negative symptoms.
Change (post training - pre training) in quality of life. | Pre Training: 3-4 days before training start. Post Training: 3-4 days after completion of training.
  World Health Organization Quality of Life Questionnaire, short version (WHOQOL-BREF). Four major domains are assessed: physical, psychological, social relationships and environment. It consists of 26 items and a maximum score of 130. Higher scores indicate a higher quality of life.
Change (follow-up - pre training) in quality of life. | Pre Training: 3-4 days before training start. Post Training: 3-4 days after completion of training. And changes in follow-up sessions: 4 and 12 weeks after completion of working memory training.
  World Health Organization Quality of Life Questionnaire, short version (WHOQOL-BREF). Four major domains are assessed: physical, psychological, social relationships and environment. It consists of 26 items and a maximum score of 130. Higher scores indicate a higher quality of life
Change (post training - pre training) in subjective cognitive capacity. | Pre Training: 3-4 days before training start. Post Training: 3-4 days after completion of training.
  Subjective Scale to Investigate Cognition in Schizophrenia (SSTICS).Scale with 21 items, maximum score of 84, higher scores indicate more subjective cognitive impairment.
Change (follow-up - pre training) in subjective cognitive capacity. | Pre Training: 3-4 days before training start. Follow-up sessions: 4 and 12 weeks after completion of working memory training.
  Subjective Scale to Investigate Cognition in Schizophrenia (SSTICS).Scale with 21 items, maximum score of 84, higher scores indicate more subjective cognitive impairment.
Differences in EEG signatures between interventional arms. | Pre Training: 3-4 days before training start. Post Training: 3-4 days after completion of training
  resting state connectivity, event-related potentials (ERP), 32-channel EEG

OTHER OUTCOMES:
Influence of genetic constitution on tDCS effectiveness | Pre Training: 3-4 days before training start
  Examination of gene polymorphisms (BDNF Val66Met, COMT Val108Met158; CACNA1C) via polymerase chain reaction (PCR).
Influence of age on tDCS effectiveness | Pre Training: 3-4 days before training start
  Age in years; demographic questionnaire
Influence of sex on tDCS effectiveness | Pre Training: 3-4 days before training start
  Sex: male, female, not specified; self report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andreas J Fallgatter, M.D., Study Director — University Hospital Tuebingen, Department of Psychiatry
Locations (2):
- Germany (2):
  - Department of Psychiatry and Psychotherapy at the Heinrich-Heine-University Duesseldorf, Düsseldorf, North Rhine-Westphalia
  - University Hospital Tuebigen, Department of Psychiatry and Psychotherapy, Tübingen

IPD SHARING:
Plan to Share IPD: Undecided